CLINICAL TRIAL: NCT01939236
Title: Traditional Chinese Medicine for Treatment of Chronic Heart Failure: A Multicenter Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Traditional Chinese Medicine for Treatment of Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Wuhan Hospital of Traditional Chinese Medicine (Other); Zhengzhou Hospital of Traditional Chinese Medicine (Other); Changchun University of Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Yichang Hospital of Traditional Chinese Medicine (Other); Dongzhimen Hospital, Beijing (Other); Guang'an Men Hospital Affiliated to China Academy of Chinese Medicine Sciences (Unknown)
Responsible Party: Principal Investigator, Wei Wang, Vice-President, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUCMlltllt1984
Record Dates: First submitted 2013-08-13; First posted 2013-09-11 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; traditional Chinese medicine; syndrome differentiation
MeSH Terms: interventions — Medicine, Chinese Traditional; Honghua extract, Carthamus tinctorius

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional Chinese medicine (Experimental): Subjects were treated with TCM 2 times per day for 28 days according to syndrome differentiation. For example, the syndrome of one patient with chronic heart failure is qi deficiency and blood stasis. He will take drug of qi deficiency and blood stasis 2 times per day for 28 days.
  Interventions: Drug: traditional Chinese medicine
- placebo (gummeline) (Placebo Comparator): Subjects were treated with placebo 2 times per day for 28 days according to syndrome differentiation. For example, the syndrome of one patient with chronic heart failure is qi deficiency and blood stasis. He will take drug of qi deficiency and blood stasis 2 times per day for 28 days.
  Interventions: Drug: Placebo (gummeline)

INTERVENTIONS:
Drug: traditional Chinese medicine — 1 bag of drug 2 times per day for 28 days according to syndrome differentiation. For example, the syndrome of one patient is qi deficiency and blood stasis, he will take drugs of qi deficiency and blood stasis each bag 2 times per day for 28days.
  Other Names: Qi deficiency：huangqi, dangshen; Blood stasis: danshen, chishao,taoren, honghua; Water retention: zexie, zhuling, cheqianzi, tinglizi; Yang deficiency: rougui, zhifuzi
  Arms: traditional Chinese medicine
Drug: Placebo (gummeline) — Placebo of each syndrome differentiation has the same weight and smell as traditional Chinese medicine of corresponding syndrome differentiation.
  1 bag of drug 2 times per day for 28 days according to syndrome differentiation.
  For example, the syndrome of one patient is qi deficiency and blood stasis, he will take drugs of qi deficiency and blood stasis each bag 2 times per day for 28 days.
  Other Names: Qi deficiency： gummeline; Blood stasis: gummeline; Water retention: gummeline; Yang deficiency: gummeline
  Arms: placebo (gummeline)

SUMMARY:
The purpose of this study is to determine whether traditional Chinese medicine as complementary treatment is safe and effective in the treatment of chronic heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) can be defined as an abnormality of cardiac structure or function leading to failure of heart to deliver oxygen at a rate commensurate with the requirements of the metabolizing tissues, despite normal filling pressures (or only at the expense of increased filling pressures). And according to the nature of the clinical presentation, HF is divided into acute or chronic HF.

In 2003, a random sample survey of 15,518 urban or rural residents between 35 and 74 years old was made in China: the prevalence rate of heart failure was 0.9%, and according to the result, there was about 4,000,000 HF subjects in China.

In China, the integrative treatment of western and traditional Chinese medicine (TCM) for HF is common and has been developed as a treatment model. TCM has been used in China and other south and east Asia countries for thousands of years. Syndrome differentiation and treatment variation are the basic principles in understanding and treatment of diseases. Investigators would like to test the hypothesis that it is efficacy and safety for patients to take TCM granules according to syndrome differentiation.

The specific aims for the study were to evaluate the efficacy and safety of TCM in treating chronic heart failure (CHF).

ELIGIBILITY:
Inclusion Criteria:

* The basic primary heart disease is coronary heart disease ( with diagnosis for coronary heart disease : confirmed by coronary angiography; confirmed by coronary CT; history of acute myocardial infarction; limb-salvage Q wave for ECG; ecg ECG test and radionuclide examination support, etc.); no history of hypertension or taking antihypertensive drugs, with blood pressure under 160/100 mmHg.
* With a history of coronary heart disease, symptoms and signs; with difficult breathing, fatigue and fluid retention (edema); with left ventricular enlargement, end systolic volume of left ventricular increase and left ventricular ejection fraction (LVEF) ≤ 40; with New York Heart Association (NYHA) functional classificationⅡ or Ⅲ.
* Male or female subjects between 40 and 75 years old;

Exclusion Criteria:

* Serious valvular heart disease, pericardial disease, cardiomyopathy, congenital heart disease, acute myocardial infarction ( within 4 weeks), cardiac shock, acute myocarditis or serious arrhythmia with the variation of hemodynamics.
* Pulmonary artery hypertension caused by pulmonary heart disease, acute or chronic pulmonary embolism, or stroke within a half year.
* Serious hepatic insufficiency ( the index of liver function being 2 times of normal one), renal insufficiency (Ccr>20%, Scr>3mg/dl or 265 μmol/L), diseases of blood system, malignant tumor, diabetes mellitus with serious complications, hyperthyroid or hypothyroid.
* Infection: fever; the numeration of leukocyte being more than 10×109/L, the percentage of neutrophile granulocyte being more than 85%; patchy shadows in X ray of Chest, meeting one of the above three.
* Pregnancy or lactation; mental disease and infectious disease patients.
* Take part in other trials within two months.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 14 days, 28 days
  The level of left ventricular ejection fraction was detected with the modified Simpson's rule at baseline and 28 days.

SECONDARY OUTCOMES:
Traditional Chinese medicine syndrome scores (TCM-SS) | 14 days, 28 days
  Before the study, all investigators took standardized training and conformance testing. Syndrome differentiation and syndrome scores were took by 3 investigators together, and the results needed to obtain two or more investigators' consent. There were 65 clinical symptoms evaluated as TCM symptoms, which was defined as TCM syndrome score. The standard of TCM symptoms scored as without 0; very light 1; light 2; medium 3; heavy 4; very heavy 5 points.
New York Heart Association (NYHA) functional classification | 14 days, 28 days
6-minute walk test (6MWT) | 14 days, 28 days
  6MWT was took according to the guidelines for the 6MWT promulgated by the American Thoracic Society at baseline and 28 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Study Chair — Beijing University of Chinese Medicine; Peng Zhang, Doctor, Principal Investigator — Wuhan Hospital of Chinese Medicine; Huihui Zhao, Doctor, Study Director — Beijing University of Chinese Medicine; Liangtao Luo, Master, Principal Investigator — Beijing University of Chinese Medicine
Locations (1):
- Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gao K, Zhao H, Gao J, Wen B, Jia C, Wang Z, Zhang F, Wang J, Xie H, Wang J, Wang W, Chen J. Mechanism of Chinese Medicine Herbs Effects on Chronic Heart Failure Based on Metabolic Profiling. Front Pharmacol. 2017 Nov 22;8:864. doi: 10.3389/fphar.2017.00864. eCollection 2017. PMID 29213243
- [Derived] Luo L, Chen J, Guo S, Wang J, Gao K, Zhang P, Chen C, Zhao H, Wang W. Chinese Herbal Medicine in the Treatment of Chronic Heart Failure: Three-Stage Study Protocol for a Randomized Controlled Trial. Evid Based Complement Alternat Med. 2015;2015:927160. doi: 10.1155/2015/927160. Epub 2015 May 18. PMID 26089951